CLINICAL TRIAL: NCT05744440
Title: Early Clinical Study of Allogenic NK Cells (JD002) in Combination With Chemotherapy in the Treatment of Relapsed or Refractory(r/r) Acute Myeloid Leukemia(AML) After Allo-HSCT
Brief Title: Safety and Efficacy of Allogenic NK Cells in Combination With Chemotherapy in the Treatment of r/r AML After Allo-HSCT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Principal Investigator, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL282-01
Record Dates: First submitted 2023-02-11; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; allogenic NK cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogenic NK cells (Experimental): Enrolled patients will receive prespecified dose of allogenic NK cells
  Interventions: Drug: allogenic NK cells

INTERVENTIONS:
Drug: allogenic NK cells — The relapsed/refractory AML after allo-HSCT patients will receive allogenic NK cells infusion up to 2 dose levels (1x10^7/kg, 5x10^7/kg) after chemotherapy with azacitidine

SUMMARY:
This is an open label, single-arm, Phase I study to evaluate the efficacy and safety of allogenic natural killer(NK) cells in subjects with refractory or relapsed AML after allogeneic hematopoietic stem cell transplantation(allo-HSCT). A leukapheresis procedure will be performed to manufacture NK cells. Prior to allogenic NK cells infusion subjects will receive chemotherapy with azacitidine.

DETAILED DESCRIPTION:
This open label, single-arm, Phase I study aims to evaluate the efficacy and safety of allogenic NK cells in subjects with refractory or relapsed AML after allo-HSCT. A leukapheresis procedure will be performed to manufacture NK cells. Prior to allogenic cells infusion subjects will receive chemotherapy with azacitidine. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable dose(MTD) and recommended phase 2 dose(rp2d) were confirmed. To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-75years old, no gender or race;
2. Expected survival is more than 3 months;
3. Eastern Cooperative Oncology Group (ECOG) score 0-2 points;
4. Diagnosed as AML in accordance with the criteria from Chinese guidelines for the diagnosis and treatment of adult AML (not acute promyelocytic leukemia (APL))(2021) and The new edition of the 2016 World Health Organization (WHO) classification system for tumors of the hematopoietic and lymphoid tissues;
5. Diagnosed as relapsed AML;
6. Measurable lesions meets at least one of the following requirements during screening: (1) Persistent positive MRD or relapse with positive minimal residual disease (MRD) in the bone marrow(BM); (2) Appearance of leukemic blasts in the peripheral blood; (3) ≥5% blasts in the BM; (4) extramedullary relapse;
7. Within 3 days prior to initial treatment, the organ functions meet the following requirements: (1) complete blood cell count: a. Absolute neutrophil counts ≥1.0×109/L and not treated with granulocyte colony stimulating factor(G-CSF) within 7 days; b.Hemoglobin ≥6g/dL(red blood cell; transfusion are permitted); c.Platelet ≥50×109/L(platelet transfusion are permitted); (2) Liver function: alanine transaminase (ALT)/ aspartate aminotransferase(AST) ≤ 3× times upper normal limit(ULN), total bilirubin ≤ 2 times ULN (direct bilirubin ≥ 1.5 times ULN is acceptable for subjects with Gilbert-Meulengracht syndrome); (3)Coagulation function: International standardized ratio (INR) or activated partial thrombin time (APTT) ≤1.5 times ULN; (4)Renal function: serum creatinine≤1.5×ULN or creatinine clearance rate ≥30ml/min; (5)Corrected serum calcium ≤14mg/dL (≤3.5mmol/L) or free calcium ≥6.5mg/dL(≥1.6mmol/L); (6)Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%;
8. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Confirmed APL;
2. ≥2 grade persistent nonhematologic toxicity of associated with prior treatment;
3. Patients with grade II-IV graft-versus-host disease (GVHD) requiring the use of immunosuppressive agents ;
4. Systemic steroid therapy exceeding the equivalent of ≥30mg/kg/day of prednisone within 48 hours prior to the first dose of study drug or other immunosuppressive therapies (except for topical and inhaled glucocorticoid therapy, or short-term prophylactic therapy with glucocorticoid) ;
5. Severe cardiovascular and cerebrovascular diseases, including: (1) Some cardiovascular and cerebrovascular diseases (such as congestive heart failure, acute myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism, etc.) occur within 6 months prior to the first dose of study drug; (2)New York Heart Association (NYHA) Class ≥3 or uncontrolled malignant arrhythmias; (3)The researchers assessed that the subjects with other cardiovascular and cerebrovascular diseases are not suitable for the study;
6. Any active infection requiring systemic therapy by intravenous infusion within 14 days prior to the first dose of study drug, including: hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), syphilis infection, or active pulmonary tuberculosis;
7. History of hypersensitivity reactions to murine protein-containing products, or macromolecular biopharmaceuticals such as antibodies or cytokines;
8. Previous or next organ transplant (except for HCT);
9. Women who are pregnant (urine/blood pregnancy test positive) or lactating;
10. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 6 months after enrollment;
11. Any unstable condition potentially imperiling patient safety and compliance;
12. Known alcohol dependence or drug dependence;
13. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 1 month
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Objective Response Rate(ORR) | 3 months
  Assessment of ORR (ORR = complete response(CR) + CRi（CR incomplete blood count recovery）+ PR(partial response)) at 3 months of treatment

SECONDARY OUTCOMES:
Progression free survival(PFS) Assessment of PFS at month 6,12 Progression free survival(PFS) | Month 6,12
  Assessment of PFS at month 6,12
Overall Survival(OS) | Month 6, 12, 18 and 24
  Assessment of OS at month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, M.D., Ph.D., Principal Investigator — Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China